CLINICAL TRIAL: NCT01383486
Title: A Pilot Self Selection Trial of an Extended-Release Over-the-Counter Analgesic
Brief Title: Self Selection Trial of Naproxen Sodium
Acronym: KEIFER SST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 15833; 2014-005305-20 (EudraCT Number)
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-06

CONDITIONS: Pain
Keywords: Self Selection Tria
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Naproxen Sodium ER (BAYH6689) or Advil IR (Experimental): Eligible subjects were provided with 24 Advil immediate-release (IR) caplets containing 200 mg Ibuprofen and Naproxen Sodium extended release (ER) tablets containing 660 mg Naproxen Sodium. Upon a single incidence of pain, subjects were instructed to review both packages and choose one product to use. Subject were not offered any additional instructions for use beyond what is on the packages.
  Interventions: Drug: Naproxen sodium ER (BAYH6689); Drug: Advil

INTERVENTIONS:
Drug: Naproxen sodium ER (BAYH6689) — Naproxen Sodium ER (BAYH6689): oral tablet upon incidence of pain
Drug: Advil — Commercially available Advil; oral caplet upon incidence of pain

SUMMARY:
A pilot trial to demonstrate that consumers can appropriately select Aleve 24 Hour for their own use based on expected duration of pain greater than 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age
* Report taking at least one dose of Over-the-counter (OTC) analgesic for pain in the past month
* Able to read and understand English
* Provide written informed consent (subjects 12-17 years of age provide written assent and/or parent or legal guardian provide written consent)
* Provide contact information

Exclusion Criteria:

* Have participated in a trial involving OTC analgesics in the last 6 months
* They or someone else in the household work for a market research company, an advertising agency, a public relations firm, a pharmaceutical company, as a healthcare professional, or as part of a health care practice (eliminated for reasons of confidentiality or increased awareness of drugs and their labels)
* Have a history of known allergies to Nonsteroidal Antiinflammatory Drugs (NSAIDs) (i.e., naproxen, ibuprofen, acetaminophen, aspirin, etc.)
* Have a history of heart surgery in the last 60 days or plans for heart surgery in the next 60 days
* Female subjects who have a positive urine pregnancy test or who are breastfeeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- United States (10):
  - Anaheim, California
  - Yorba Linda, California
  - Pembroke Pines, Florida
  - Griffin, Georgia
  - Andover, Minnesota
  - Roseville, Minnesota
  - Bountiful, Utah
  - West Jordan, Utah
  - Bellevue, Washington
  - Seattle, Washington

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 435 subjects were screened, 384 were qualified for participation, 259 subjects presented at pharmacy to begin enrollment procedures, 254 gave inform consent, 1 subject refused to give pregnancy test, so 253 subject received the investigational products.
Groups:
- Naproxen Sodium ER (BAY H6689) or Advil IR: Eligible subjects were provided with 24 Advil immediate-release (IR) caplets containing 200 mg Ibuprofen and 20 Aleve 24 Hour extended release (ER) tablets containing 660 mg Naproxen Sodium. Upon a single incidence of pain, subjects were instructed to review both packages and choose one product to use. Subject were not offered any additional instructions for use beyond what is on the packages.
Period: Overall Study
Arm/Group | Naproxen Sodium ER (BAY H6689) or Advil IR
Started | 253 (Number of participants who were provided with investigational products)
Treated | 237 (Number of participants who took any study medication (Safety Population))
Completed | 235 (Took any study medication and gave estimated duration of pain (Selection Evaluation Population))
Not Completed | 18
Not completed — Lost to Follow-up | 10
Not completed — Incomplete information for analysis | 2
Not completed — Did not take any product | 6

BASELINE CHARACTERISTICS:
Arm/Group | Naproxen Sodium ER (BAY H6689) or Advil IR
Number analyzed (Participants) | 235
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (14.3)
Gender [Number; unit: Participants] — 119 females; 115 males; 1 subject refused to provide gender information
  Participants
    Female | 119
    Male | 115

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Selected Naproxen Sodium ER and Expected Their Pain to Last More Than 12 Hours
Description: Participants were instructed to select a product for use upon their pain episode and then call a toll-free number for an interview within 30 minutes of the selection decision. Participants who did not call were interviewed after 14 days for data collection. The primary endpoint was derived from 2 variables: 1) number of participants who selected Naproxen Sodium ER and reported expected duration of pain less than or equal to 12 hrs (A); 2) number of participants who selected Naproxen Sodium ER and report expected duration of pain greater than 12 hrs (B). The results was calculated as B/(A+B).
Time Frame: up to 14 days
Population: Only subjects who chose naproxen sodium were included in the analysis.
Measure: Number; unit: Percentage of participants
Groups:
- Naproxen Sodium ER (BAY H6689) or Advil IR: Eligible subjects were provided with 24 Advil immediate-release (IR) caplets containing 200 mg Ibuprofen and Naproxen Sodium extended release (ER) tablets containing 660 mg Naproxen Sodium. Upon a single incidence of pain, subjects were instructed to review both packages and choose one product to use. Subject were not offered any additional instructions for use beyond what is on the packages.
Arm/Group | Naproxen Sodium ER (BAY H6689) or Advil IR
Number analyzed (Participants) | 182
Percentage of participants | 72.0 [64.9 to 78.4]

2. Secondary Outcome: The Percentage of Participants Who Selected Naproxen Sodium ER , Expected Their Pain to Last More Than 12 Hours and Reported Their Selection Decision Within First 24 Hours
Time Frame: Within 24 hours of their selection decision taken up to 14 days
Population: Subgroup of Selection Evaluation Population
Measure: Number; unit: Percentage of participants
Groups:
- Naproxen Sodium ER (BAY H6689) or Advil IR: Eligible subjects were provided with 24 Advil IR caplets containing 200 mg Ibuprofen and Naproxen Sodium extended release (ER) tablets containing 660 mg Naproxen Sodium. Upon a single incidence of pain, subjects were instructed to review both packages and choose one product to use. Subject were not offered any additional instructions for use beyond what is on the packages.
Arm/Group | Naproxen Sodium ER (BAY H6689) or Advil IR
Number analyzed (Participants) | 151
Percentage of participants | 71.5 [63.6 to 78.6]

3. Secondary Outcome: The Percentage of Low Literacy Participants Who Selected Naproxen Sodium ER and Expected Their Pain to Last More Than 12 Hours
Description: In addition to the primary outcome measure evaluated for all selection evaluable participants, this secondary outcome was evaluated separately for low literacy participants. Low Literacy Participants are defined as those who had REALM (Rapid Estimate of Adult Literacy in Medicine) score </= 60 at visit 1.
Time Frame: Up to 14 days
Population: Subgroup of Selection Evaluation Population: low literacy participants who had REALM score </= 60 at visit 1 and chose naproxen sodium.
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium ER (BAY H6689) or Advil IR
Number analyzed (Participants) | 31
Percentage of participants | 64.5 [45.4 to 80.8]

ADVERSE EVENTS:
Arm/Group | Naproxen Sodium ER (BAY H6689) or Advil IR
Serious Adverse Events (participants affected / at risk) | 0/237
Other Adverse Events (participants affected / at risk) | 14/237
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium ER (BAY H6689) or Advil IR (N=237)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Pain in extremity (General disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasopharyngtis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days